CLINICAL TRIAL: NCT04216290
Title: Phase II Study of Bladder-SparIng ChemoradiatioN With Durvalumab in Clinical Stage III, Node PosItive BladdeR CancEr (INSPIRE)
Brief Title: A Study of Chemotherapy and Radiation Therapy Compared to Chemotherapy and Radiation Therapy Plus MEDI4736 (Durvalumab) Immunotherapy for Bladder Cancer Which Has Spread to the Lymph Nodes, INSPIRE Trial
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2019-08628; NCI-2019-08628 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EA8185 (Other: ECOG-ACRIN Cancer Research Group); EA8185 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2019-12-31; First posted 2020-01-02 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Bladder Urothelial Carcinoma; Stage III Bladder Cancer AJCC v8
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Specimen Handling; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Cystoscopy; durvalumab; Immunoglobulin G; Disulfides; Fluorouracil; dehydroftorafur; Gemcitabine; Magnetic Resonance Spectroscopy; Mitomycin; Mitozytrex; Watchful Waiting; Observation; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Step 1, Arm C (durvalumab, radiation therapy, chemotherapy) (Experimental): Patients undergo radiation therapy for 6.5-8 weeks. Beginning 4 days before or after starting radiation therapy, patients receive durvalumab IV over 60 minutes on day 1 of each cycle. Treatment repeats every 21 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Beginning 4 days before or after starting radiation therapy, patients also receive gemcitabine hydrochloride IV over 30-60 minutes BIW for 6 weeks; or cisplatin IV over 30-60 minutes QW for 6 weeks; or mitomycin IV over 30 minutes on day 1 of radiation and fluorouracil IV continuous infusion on days 1-5 and 16-20 of radiation in the absence of disease progression or unacceptable toxicity. Patients also undergo bladder biopsy on study, cystoscopy on study and during follow-up, as well as CT or MRI throughout the trial. Patients may also undergo tumor tissue and blood sample collection on study.
  Interventions: Procedure: Biopsy of Bladder; Procedure: Biospecimen Collection; Drug: Cisplatin; Procedure: Computed Tomography; Procedure: Cystoscopy; Biological: Durvalumab; Drug: Fluorouracil; Drug: Gemcitabine Hydrochloride; Procedure: Magnetic Resonance Imaging; Drug: Mitomycin; Radiation: Radiation Therapy
- Step 1, Arm D (radiation therapy, chemotherapy) (Active Comparator): Patients undergo radiation therapy for 6.5-8 weeks. Beginning 4 days before or after starting radiation therapy, patients also receive gemcitabine hydrochloride IV over 30-60 minutes BIW for 6 weeks; or cisplatin IV over 30-60 minutes QW for 6 weeks; or mitomycin IV over 30 minutes on day 1 of radiation and fluorouracil IV continuous infusion on days 1-5 and 16-20 of radiation in the absence of disease progression or unacceptable toxicity. Patients also undergo bladder biopsy on study, cystoscopy on study and during follow-up, as well as CT or MRI throughout the trial. Patients may also undergo tumor tissue and blood sample collection on study.
  Interventions: Procedure: Biopsy of Bladder; Procedure: Biospecimen Collection; Drug: Cisplatin; Procedure: Computed Tomography; Procedure: Cystoscopy; Drug: Fluorouracil; Drug: Gemcitabine Hydrochloride; Procedure: Magnetic Resonance Imaging; Drug: Mitomycin; Radiation: Radiation Therapy
- Step 2, Arm E (durvalumab) (Experimental): Patients previously randomized to Arm C (chemoradiation and durvalumab) who achieve clinical CR or clinical benefit receive durvalumab IV over 60 minutes on day 1 of each cycle. Treatment repeats every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo bladder biopsy on study, cystoscopy on study and during follow-up, as well as CT or MRI throughout the trial. Patients may also undergo tumor tissue and blood sample collection on study.
  Interventions: Procedure: Biopsy of Bladder; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Cystoscopy; Biological: Durvalumab; Procedure: Magnetic Resonance Imaging
- Step 2, Arm F (observation) (Active Comparator): Patients previously randomized to Arm D (chemoradiation) who achieve clinical CR or clinical benefit undergo observation undergo observation. Patients also undergo bladder biopsy on study, cystoscopy on study and during follow-up, as well as CT or MRI throughout the trial. Patients may also undergo tumor tissue and blood sample collection on study.
  Interventions: Procedure: Biopsy of Bladder; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Cystoscopy; Procedure: Magnetic Resonance Imaging; Other: Patient Observation

INTERVENTIONS:
Procedure: Biopsy of Bladder — Undergo bladder biopsy
  Other Names: Bladder Biopsy
Procedure: Biospecimen Collection — Undergo tumor tissue and blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
  Arms: Step 1, Arm C (durvalumab, radiation therapy, chemotherapy); Step 1, Arm D (radiation therapy, chemotherapy)
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Cystoscopy — Undergo cystoscopy
  Other Names: CS
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI 4736; MEDI-4736; MEDI4736
  Arms: Step 1, Arm C (durvalumab, radiation therapy, chemotherapy); Step 2, Arm E (durvalumab)
Drug: Fluorouracil — Given IV
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
  Arms: Step 1, Arm C (durvalumab, radiation therapy, chemotherapy); Step 1, Arm D (radiation therapy, chemotherapy)
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; Gemcitabine HCI; Gemzar; LY 188011; LY-188011; LY188011
  Arms: Step 1, Arm C (durvalumab, radiation therapy, chemotherapy); Step 1, Arm D (radiation therapy, chemotherapy)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Mitomycin — Given IV
  Other Names: Ametycine; Jelmyto; MITO; Mito-C; Mito-Medac; Mitocin; Mitocin-C; Mitolem; Mitomycin C; Mitomycin pyelocalyceal; Mitomycin-C; Mitomycin-X; Mitomycine C; Mitosol; Mitozytrex; Mutamycin; Mutamycine; NCI-C04706
  Arms: Step 1, Arm C (durvalumab, radiation therapy, chemotherapy); Step 1, Arm D (radiation therapy, chemotherapy)
Other: Patient Observation — Undergo observation
  Other Names: Active Surveillance; deferred therapy; expectant management; Observation; Watchful Waiting
  Arms: Step 2, Arm F (observation)
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
  Arms: Step 1, Arm C (durvalumab, radiation therapy, chemotherapy); Step 1, Arm D (radiation therapy, chemotherapy)

SUMMARY:
This phase II trial studies the benefit of adding an immunotherapy drug called MEDI4736 (durvalumab) to standard chemotherapy and radiation therapy in treating bladder cancer which has spread to the lymph nodes. Drugs used in standard chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Cisplatin is in a class of medications known as platinum-containing compounds. It works by killing, stopping or slowing the growth of tumor cells. Radiation therapy uses high-energy x-rays to kill tumor cells and shrink tumors. Immunotherapy with durvalumab may help the body's immune system attack the cancer and may interfere with the ability of tumor cells to grow and spread. Giving chemotherapy and radiation therapy with the addition of durvalumab may work better in helping tumors respond to treatment compared to chemotherapy and radiation therapy alone. Patients with limited regional lymph node involvement may benefit from attempt at bladder preservation, and use of immunotherapy and systemic chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the clinical complete response rate (cCR) after chemoradiotherapy (chemoRT) with or without durvalumab in node-positive bladder cancer patients.

SECONDARY OBJECTIVES:

I. To compare the toxicity profile in both arms using the Common Terminology Criteria for Adverse Events (CTCAE).

II. To estimate the progression-free survival (PFS) in both arms. III. To estimate overall survival (OS) post randomization in both arms. IV. To estimate the bladder intact event free survival (BIEFS) in both arms. V. To estimate the metastasis free survival (MFS) in both arms. VI. To estimate bladder cancer specific survival in both arms. VII. To estimate the complete clinical response duration in both arms. VIII. To estimate salvage cystectomy rates in both arms.

EXPLORATORY OBJECTIVE:

I. Planned subgroup analyses for clinical outcome (clinical complete response [CR] rate post chemoRT +/- durvalumab, MFS, OS, PFS) based on stratification factors.

TRANSLATIONAL OBJECTIVE:

I. To collect and bank tumor tissue and blood specimens at pre-and post-treatment with chemoRT +/- durvalumab to determine predictive or prognostic markers.

OUTLINE:

STEP 1 - Randomization: Patients are randomized to 1 of 2 arms.

ARM C: Patients undergo radiation therapy for 6.5-8 weeks. Beginning 4 days before or after starting radiation therapy, patients receive durvalumab intravenously (IV) over 60 minutes on day 1 of each cycle. Treatment repeats every 21 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Beginning 4 days before or after starting radiation therapy, patients also receive gemcitabine hydrochloride IV over 30-60 minutes twice a week (BIW) for 6 weeks; or cisplatin IV over 30-60 minutes once a week (QW) for 6 weeks; or mitomycin IV over 30 minutes on day 1 of radiation and fluorouracil IV continuous infusion on days 1-5 and 16-20 of radiation in the absence of disease progression or unacceptable toxicity. Patients also undergo bladder biopsy on study, cystoscopy on study and during follow-up, as well as computed tomography (CT) or magnetic resonance imaging (MRI) throughout the trial. Patients may also undergo tumor tissue and blood sample collection on study.

ARM D: Patients undergo radiation therapy for 6.5-8 weeks. Beginning 4 days before or after starting radiation therapy, patients also receive gemcitabine hydrochloride IV over 30-60 minutes BIW for 6 weeks; or cisplatin IV over 30-60 minutes QW for 6 weeks; or mitomycin IV over 30 minutes on day 1 of radiation and fluorouracil IV continuous infusion on days 1-5 and 16-20 of radiation in the absence of disease progression or unacceptable toxicity. Patients also undergo bladder biopsy on study, cystoscopy on study and during follow-up, as well as CT or MRI throughout the trial. Patients may also undergo tumor tissue and blood sample collection on study.

STEP 2 - Registration: Patients are assigned to 1 of 2 arms.

ARM E: Patients previously randomized to Arm C (chemoradiation and durvalumab) who achieve clinical CR or clinical benefit receive durvalumab IV over 60 minutes on day 1 of each cycle. Treatment repeats every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo bladder biopsy on study, cystoscopy on study and during follow-up, as well as CT or MRI throughout the trial. Patients may also undergo tumor tissue and blood sample collection on study.

ARM F: Patients previously randomized to Arm D (chemoradiation) who achieve clinical CR or clinical benefit undergo observation. Patients also undergo bladder biopsy on study, cystoscopy on study and during follow-up, as well as CT or MRI throughout the trial. Patients may also undergo tumor tissue and blood sample collection on study.

After completion of study treatment, patients are followed up every 12 weeks for 1 year, every 6 months for year 2, and then annually for years 3-4.

ELIGIBILITY:
Inclusion Criteria:

* STEP 1 (RANDOMIZATION) ELIGIBILITY CRITERIA:
* Patient must be >= 18 years of age.
* Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 at the time of step 1 randomization.
* Patient must have histologically proven pure or mixed urothelial cancer of the bladder.

  * NOTE: Small cell carcinoma is excluded, however other variant histologies are permitted provided a component of urothelial carcinoma is present.
* Patient must have documented node-positive and non-metastatic disease (any T, any N, M0). Node positivity must have been defined prior to receiving any systemic chemotherapy or induction chemotherapy.

Node positivity can fall into either of the following categories and will be defined by imaging and/or biopsy:

* A lymph node >= 1.0 cm in short axis on imaging (i.e., CT or MRI or positron emission tomography [PET]/CT).
* A lymph node that is < 1 cm on imaging with either a biopsy confirming involvement with cancer or high suspicion of cancer.

  * For patients who have received induction chemotherapy (any type of systemic chemotherapy) for node positive bladder cancer prior to enrollment, there must be no signs of disease progression (CR/partial response [PR] or stable disease [SD]) based on restaging imaging and cystoscopy, which consists of:
* CT chest, abdomen, and pelvis obtained after completion of induction chemotherapy and within 8 weeks prior to step 1 randomization.

  * NOTE: MRI can be used instead of CT per treating physician discretion.
* Cystoscopic evaluation and attempt to perform maximal transurethral resection of bladder tumor (TURBT) performed by the participating urologist after completion of induction chemotherapy and within 12 weeks prior to step 1 randomization. If maximal TURBT is not possible for medical reasons, the enrollment must be discussed and approved with the study chair. Documentation of correspondences with the study chair must be kept on file.
* Patients who achieve CR upon cystoscopy per urologist with no visible tumor (i.e., no need for additional TURBT), are allowed to proceed in the study as adequate resection with no residual disease in bladder.

  * For patients who have did not receive induction chemotherapy (any type of systemic chemotherapy) for node positive bladder cancer prior to enrollment, the following must be obtained:
* CT chest, abdomen, and pelvis completed within 8 weeks prior to step 1 randomization.

  * NOTE: MRI can be used instead of CT per treating physician discretion.
* Cystoscopic evaluation and attempt to perform maximal TURBT performed by the participating urologist within 12 weeks prior to step 1 randomization. If maximal TURBT is not possible for medical reasons, the enrollment must be discussed and approved with the study chair. Documentation of correspondences with the study chair must be kept on file.
* For patients who may need repeat TURBT if their old TURBT has fallen out of window: If urologist determine no visible tumor (i.e., no need for additional resection) upon cystoscopy, they are allowed to proceed in the study as complete resection.

  * Patient must not have received any previous radiation therapy to the pelvic area.
  * Patient must agree to undergo CT simulation and treatment planning. If this is the first case registered at the site, then a pre-treatment radiation therapy (RT) review will be required and will take up to 3 business days. The patient cannot start radiation treatment prior to successful completion of this pre-treatment review. Therefore, careful planning is necessary to meet the deadline of starting radiation within 20 business days of step 1 randomization.
  * Patient must not have presence of concomitant active upper tract tumors or urethra tumors. History of previously adequately treated non-muscle invasive bladder cancer (NMIBC) are eligible. Previously treated urothelial cancer or histological variant at any site outside of the urinary bladder are allowed, provided they have been Ta/T1/carcinoma in situ (CIS) and post treatment follow up imaging and endoscopic evaluation shows no evidence of disease.
  * Patients with previous exposure to immune checkpoint inhibitor for non-muscle invasive disease are eligible. If given for NMIBC, the last dose must have been completed > 12 months prior to step 1 randomization.
  * Patient must not be pregnant or breast-feeding due to the potential harm to an unborn fetus and possible risk for adverse events in nursing infants with the treatment regimens being used.

All patients of childbearing potential must have a blood test or urine study within 14 days prior to step 1 randomization to rule out pregnancy.

A patient of childbearing potential is defined as any patient, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy; or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).

* Patients must not expect to conceive or father children by using accepted and effected method(s) of contraception or by abstaining from sexual intercourse from the time of step 1 randomization for the duration of their participation in the study and continue for at least 3 months after the last dose of protocol treatment.
* Leukocytes >= 3,000/mcL (obtained < 14 days prior to step 1 randomization).
* Absolute neutrophil count (ANC) >= 1,500/mcL (obtained < 14 days prior to step 1 randomization).
* Hemoglobin >= 9 g/dL (obtained < 14 days prior to step 1 randomization).
* Platelets >= 100,000/mcL (obtained < 14 days prior to step 1 randomization).
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (obtained < 14 days prior to step 1 randomization).
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional ULN (obtained < 14 days prior to step 1 randomization).
* Adequate renal function as evidenced by calculated (Cockcroft's formula) creatinine clearance or 24 hours actual creatinine clearance >= 30mL/min. The creatinine used to calculate the clearance result must have been obtained within 14 days prior to step 1 randomization. Actual body weight, not ideal body weight, must be used in the calculation.
* Patients with human immunodeficiency virus (HIV) on effective anti-retroviral therapy with undetectable viral load within 6 months of step 1 randomization are eligible for this trial.
* For patients with autoimmune conditions, patient must not have history of prior documented autoimmune disease within 2 years prior to step 1 randomization.

  * NOTE: Patient with vitiligo, Grave's disease, eczema or psoriasis (not requiring systemic treatment within 2 years prior to step 1 randomization) are not excluded. Patients with history of completely resolved childhood asthma or atopy are not excluded. Patients with asthma not requiring more than 10 mg/d or equivalent of prednisone are not excluded. Patients with well-controlled hypothyroidism on thyroxine replacement will be eligible as well. Patients with known history of hypoadrenalism on maintenance steroids will be eligible. Patients with type I diabetes mellitus will be eligible, provided their disease is well controlled. History of autoimmune related alopecia is also not an exclusion criteria.
  * Patient with active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis) are not eligible.
  * Patient with a history of and/or confirmed pneumonitis are not eligible.
  * Patient with a history of primary immunodeficiency are not eligible.
  * Patient with history of allogeneic organ transplant are not eligible.
* Patient must not have an active infection, including:

  * Tuberculosis (based on clinical evaluation that includes clinical history, physical examination, and radiographic findings, and tuberculosis testing in line with local practice).
  * Hepatitis B (known positive hepatitis B virus [HBV] surface antigen [HBsAg] result). Past or resolved HBV infection (defined as the presence of hepatitis b core antibody [anti-HBc] and absence of HBsAg) are eligible.
  * Hepatitis C. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction test is negative for HCV ribonucleic acid (RNA).
* Patient must not have clinically significant liver disease that precludes patient from treatment regimens prescribed on the study (including, but not limited to, active viral, alcoholic or other autoimmune hepatitis, cirrhosis or inherited liver disease).
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial. Site is encouraged to discuss with the study chair if needed prior to enrollment.
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class IIB or better.
* Patient must not have received live attenuated vaccine within 30 days prior to the first dose of durvalumab

  * NOTE: Patient, if enrolled, must not receive live vaccine whilst receiving durvalumab and up to 30 days after the last dose of durvalumab.
  * NOTE: Patient is permitted to receive inactivated vaccines and any non-live vaccines including those for the seasonal influenza and coronavirus disease 2019 (COVID-19) (Note: intranasal influenza vaccines, such as Flu-Mist (registered trademark) are live attenuated vaccines and are not allowed). If possible, it is recommended to separate study drug administration from vaccine administration by about a week (primarily in order to minimize an overlap of adverse events).
* Patient must not have current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

  * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection).
  * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent.
  * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
* Patient must not have any unresolved toxicity (National Cancer Institute [NCI] CTCAE grade >= 2) from previous anti-cancer therapy with the exception of alopecia, vitiligo, and the laboratory values.

  * NOTE: Patients with grade >= 2 neuropathy will be evaluated on a case-by-case basis after consultation with the study chair.
  * NOTE: Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the study chair. Documentation of correspondences with the study chair must be kept on file.
* STEP 2 (REGISTRACTION: ADJUVANT DURVALUMAB VERSUS [VS] OBSERVATION) ELIGIBILITY CRITERIA:
* Patient must have evaluation to determine clinical outcome post step 1 treatment (chemoRT+/- durvalumab) with imaging (CT chest, abdomen, and pelvis) (preferably contrast with urogram, if not contraindicated) and cystoscopy with biopsy confirmation to ensure no progression and absence of >= T2 disease in the bladder. Patient should be registered to step 2 within 28 days from the determination of primary response to step 1 treatment. However, for patients previously on Arm C, an additional 4 week delay to step 2 registration is allowed.
* Patient on the chemoRT+ durvalumab (Arm C) must meet the following:

  * Patient must have achieved either complete clinical response OR have demonstrated clinical benefit prior to continuing onto adjuvant durvalumab.
  * Patients who are to go on the adjuvant durvalumab (Arm E) must have recovered to at least grade 2 or less immune related adverse event (AE) prior to starting treatment except for immune related alopecia, clinically asymptomatic endocrinopathies. For patients who may have gotten immune related AEs during chemoRT+ durvalumab (Arm C), step 2 registration could be delayed up to additional 4 weeks to ensure recovery to at least grade 2 or lower prior to starting adjuvant therapy. However patients with durvalumab related AEs that require permanent discontinuation of durvalumab will not continue on the adjuvant treatment regardless of the response.
  * Patient must not have experienced immune related neurological disorder described as Guillain-Barré syndrome, myasthenic syndrome or myasthenia gravis, or meningoencephalitis during chemoRT+ durvalumab treatment.
  * Patient must not have experienced immune related myocarditis or immune related pericarditis during chemoRT+ durvalumab treatment.
  * ANC >= 1,000 mcL (must be obtained < 28 days prior to step 2 registration).
  * Hemoglobin >= 8g/dL (must be obtained < 28 days prior to step 2 registration).
  * Platelets >= 70,000 mcL (must be obtained < 28 days prior to step 2 registration).

    * NOTE: If recovery is not achieved, blood counts could be repeated weekly and step 2 registration could be delayed up to additional 4 weeks.
* Patient on the chemoRT arm (Arm D) must have achieved either complete clinical response OR have demonstrated clinical benefit prior to be placed on the observation alone arm (Arm F).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2021-03-17 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Clinical complete response (CR) | Up to 4 years
  Defined as CR in bladder and nodes with no distant metastases. This study is designed to detect an improvement in clinical CR rate from 37.5% on the chemoradiation (chemoRT) arm to 62.5% on the chemoRT + durvalumab arm. Patients who receive any chemoRT +/- durvalumab will be included in the interim and final analyses. Those who are unevaluable post chemoRT +/- durvalumab, such as those patients who drop out before completing treatment post randomization or drop out prior to evaluation of first response or those patients who cannot get computed tomography scan and or cystoscopy to evaluate for response will be considered non-responders.

SECONDARY OUTCOMES:
Metastasis-free survival | From randomization to first evidence of metastatic disease or death from any cause, assessed up to 4 years
  Patients who are alive and metastasis-free will be censored at date of last assessment. The Kaplan-Meier method will be used to estimate time-to-event endpoints and stratified Cox proportional hazards models will be used to estimate hazard ratios in all eligible patients.
Bladder-intact event-free survival (BI-EFS) | From randomization to the first BI-EFS event, assessed up to 4 years
  Events of interest are presence of muscle-invasive bladder cancer, clinical evidence of progression of nodal involvement or development of metastatic disease, radical cystectomy, or death due to any cause. Patients last known to be BI-EFS event-free will be censored at the date of last assessment. Patients alive without disease assessment will be censored at randomization. The Kaplan-Meier method will be used to estimate time-to-event endpoints and stratified Cox proportional hazards models will be used to estimate hazard ratios in all eligible patients.
Bladder cancer specific survival | From randomization to death from bladder cancer, assessed up to 4 years
  Deaths due to other causes will be considered competing events and patients known to be alive will be censored at the date of last contact. The Kaplan-Meier method will be used to estimate time-to-event endpoints and stratified Cox proportional hazards models will be used to estimate hazard ratios in all eligible patients.
Overall survival | From randomization to death from any cause, assessed up to 4 years
  Patients still alive will be censored at date of last contact. The Kaplan-Meier method will be used to estimate time-to-event endpoints and stratified Cox proportional hazards models will be used to estimate hazard ratios in all eligible patients.
Progression-free survival | From randomization to first of local progression, nodal or distant metastasis, or death from any cause, assessed up to 4 years
  Patients last known to be alive and progression-free will be censored at the date of last contact. The Kaplan-Meier method will be used to estimate time-to-event endpoints and stratified Cox proportional hazards models will be used to estimate hazard ratios in all eligible patients.
Complete response duration | From the date of the biopsy documenting the complete response to the time of muscle invasive recurrence, local progression, evidence of metastatic disease or death due to any cause, assessed up to 4 years
  Patients will be censored at the date of last disease assessment. The Kaplan-Meier method will be used to estimate time-to-event endpoints and stratified Cox proportional hazards models will be used to estimate hazard ratios in all eligible patients.
Salvage cystectomy rate | Up to 4 years
  Will be reported as a proportion of patients who do not experience clinical benefit and undergo salvage cystectomy after chemoRT +/- durvalumab along with a 90% confidence interval. The Kaplan-Meier method will be used to estimate time-to-event endpoints and stratified Cox proportional hazards models will be used to estimate hazard ratios in all eligible patients.
Incidence of adverse events | Up to 4 years
  Assessed using the Common Terminology Criteria for Adverse Events version 5.0. Toxicity will be evaluated in all treated patients, regardless of eligibility.

CONTACTS AND LOCATIONS:
Overall Officials: Monika Joshi, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (216):
- United States (216):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Edward Hines Jr VA Hospital, Hines, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - East Jefferson General Hospital, Metairie, Louisiana
  - LSU Healthcare Network / Metairie Multi-Specialty Clinic, Metairie, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - SMC Center for Hematology Oncology Union, Union, South Carolina
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Sovah Health Martinsville, Martinsville, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Welch Cancer Center, Sheridan, Wyoming

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

DOCUMENTS (1):
  • Informed Consent Form (2024-05-16): https://cdn.clinicaltrials.gov/large-docs/90/NCT04216290/ICF_000.pdf